CLINICAL TRIAL: NCT00009178
Title: Treatment of Bulimia Nervosa in a Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Walsh (completed); R01DK053635-03 (NIH)
Record Dates: First submitted 2001-01-23; First posted 2001-01-23 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Bulimia Nervosa
Keywords: Primary Care; Fluoxetine
MeSH Terms: conditions — Bulimia Nervosa | interventions — Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine
Behavioral: Guided Self-Help

SUMMARY:
Bulimia Nervosa is a frequent problem for young women. It is widely assumed that this disorder cannot be treated effectively in a primary care setting. This assumption has never been tested empirically, and is probably incorrect.

In the last 15 years, effective treatment interventions for Bulimia Nervosa have been developed and validated in specialized treatment centers. The broad aim of this proposal is to examine whether these treatments, suitably adapted, can be usefully transferred to general health care settings. Specifically, the proposed study will determine the relative and combined effectiveness of the two leading treatments for Bulimia Nervosa in a primary care setting. The two major interventions are treatment with an antidepressant medication, fluoxetine, and with a form of cognitive behavioral therapy, guided self-help, designed for use in primary care.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for bulimia nervosa with a modified frequency criterion of at least once a week

Exclusion Criteria:

* Physical disorder requiring hospitalization or ongoing treatment likely to affect eating and/or weight
* Significant suicidal ideation or behavior
* Subjects judged unable to tolerate four-month treatments available in the study because of comorbid psychiatric conditions
* Current drug or alcohol dependence
* Current anorexia nervosa
* Pregnancy or any physical condition or treatments known to influence eating and weight
* Current psychiatric treatment or medication known to affect eating or weight
* Previous course of fluoxetine at a dose of 60 mg. per day for at least four weeks
* Allergy to fluoxetine
* Previous course of cognitive behavioral therapy for Bulimia Nervosa at a qualified center

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-03; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: B. T. Walsh, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Waller D, Fairburn CG, McPherson A, Kay R, Lee A, Nowell T. Treating bulimia nervosa in primary care: a pilot study. Int J Eat Disord. 1996 Jan;19(1):99-103. doi: 10.1002/(SICI)1098-108X(199601)19:13.0.CO;2-L. PMID 8640208